CLINICAL TRIAL: NCT02418585
Title: A Randomized, Double-blind, Multicenter, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Flexible Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Subjects With Treatment-resistant Depression
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Flexible Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Participants With Treatment-resistant Depression
Acronym: TRANSFORM-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107147; ESKETINTRD3002 (Other: Janssen Research & Development, LLC); 2014-004585-22 (EudraCT Number)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Treatment-resistant Depression
Keywords: Treatment-resistant Depression; Esketamine; Placebo; Oral Antidepressant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Duloxetine Hydrochloride; Antidepressive Agents; Escitalopram; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine plus oral antidepressant (Experimental): Participants will self-administer esketamine intranasally twice per week for 4 weeks as a flexible dose regimen in the Double-Blind Induction Phase. All participants will start at a dose of 56 mg on Day 1. On Day 4, the dose may be increased to 84 mg or remain at 56 mg per investigator's discretion. On Days 8 and 11 the dose may be increased to 84 mg (from 56 mg), remain same, or be reduced to 56 mg (from 84 mg) per investigator's discretion. On Day 15, a dose reduction from 84 mg to 56 mg is permitted, if required for tolerability; no dose increase permitted. After Day 15, dose must remain stable (unchanged). In addition participants will simultaneously initiate a new, open-label oral antidepressant (duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Esketamine; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)
- Placebo plus oral antidepressant (Active Comparator): Participants will self-administer matching placebo, intranasally, twice per week for 4 weeks as a flexible dose regimen in Double-Blind Induction Phase. In addition participants will simultaneously initiate a new, open-label oral antidepressant (ie, duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1 that will be continued for the duration of Double-Blind Induction Phase.
  Interventions: Drug: Placebo; Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)

INTERVENTIONS:
Drug: Esketamine — Participants will self-administer either 56 mg or 84 mg of esketamine, intranasally, twice per week as a flexible dose regimen in the Double-Blind Induction Phase.
  Arms: Intranasal Esketamine plus oral antidepressant
Drug: Placebo — Participants will self-administer matching placebo, intranasally, twice per week for 4 weeks as a flexible dose regimen in the Double-Blind Induction Phase.
  Arms: Placebo plus oral antidepressant
Drug: Duloxetine (Oral Antidepressant) — Duloxetine could be selected as the oral antidepressant medication by the investigator based on review of Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and relevant prior antidepressant medication information. The minimum therapeutic dose is 60 milligram per day (mg/day).
Drug: Escitalopram (Oral antidepressant) — Escitalopram could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Escitalopram will be titrated upto a dose of 20 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 10 mg/day.
Drug: Sertraline (Oral Antidepressant) — Sertraline could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Sertraline will be titrated upto a dose of 150 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 50 mg/day.
Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant) — Venlafaxine Extended Release could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Venlafaxine Extended Release will be titrated upto a dose of 225 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 150 mg/day.

SUMMARY:
The purpose of this study is to compare the efficacy and safety of switching treatment-resistant depression (TRD) subjects from a prior antidepressant treatment (to which they have not responded) to either intranasal esketamine plus a new oral antidepressant or switching to a new oral antidepressant plus intranasal placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither the researchers nor the subjects know what treatment the subject is receiving), active-controlled, multicenter study (more than 1 study site) in subjects with TRD to assess the efficacy, safety, and tolerability of flexible doses of intranasal esketamine plus a newly initiated oral antidepressant compared with a newly initiated oral antidepressant (active comparator) plus intranasal placebo. The study will consist of 3 phases: Screening/Prospective Observational Phase (4-7 weeks), Double-blind Induction Phase (4-weeks), Follow-up Phase (24-weeks). Subjects who rollover into a long-term maintenance study will not participate in the Follow-up Phase. The antidepressant treatment, as well as any other ongoing medications being taken for depression at screening (including adjunctive/ augmentation therapies), will continue unchanged, at the same dosage, from the start of Week 1 through the end of Week 4 of the screening/prospective observational phase. Subjects' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form (ICF), participant must be a man or woman 18 (or older if the minimum legal age of consent in the country in which the study is taking place is greater than [>]18) to 64 years of age, inclusive
* At the start of the screening/prospective observational phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) (if single-episode MDD, the duration must be greater than or equal to [>=] 2 years) or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* At the start of the screening/prospective observational phase, participant must have an Inventory of Depressive Symptomatology-Clinician rated ( IDS-C30) total score of greater than or equal to (>=) 34
* At the start of the screening/prospective observational phase, participant must have had non-response (greater than or equal to [<=25] percent [%] improvement) to ≥1 but less than or equal to (<=) 5 (if current episode is >2 years, upper limit is applicable to only the last 2 years) oral antidepressant treatments in the current episode of depression, assessed using the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and documented by medical history and pharmacy/prescription records, for the current episode of depression. In addition, the participant is taking a different oral antidepressant treatment (on the MGH-ATRQ) for at least the previous 2 weeks at or above the minimum therapeutic dose
* The participant's current major depressive episode, depression symptom severity (Week 1 MADRS total score >=28 required), and antidepressant treatment response in the current depressive episode, must be confirmed using a Site Independent Qualification Assessment

Exclusion Criteria:

* Participants who have previously demonstrated nonresponse of depressive symptoms to esketamine or ketamine in the current major depressive episode, to all 4 of the oral antidepressant treatment options available for the double-blind induction phase (ie, duloxetine, escitalopram, sertraline, and venlafaxine extended release [XR]) in the current major depressive episode (based on MGH-ATRQ), or an adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT
* Participant has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychosis, bipolar or related disorders (confirmed by the MINI), comorbid obsessive compulsive disorder, intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening/prospective observational phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Participants with history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (48):
- United States (10):
  - Birmingham, Alabama
  - Orange, California
  - San Rafael, California
  - Maitland, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Gaithersburg, Maryland
  - Boston, Massachusetts
  - Philadelphia, Pennsylvania
  - Dallas, Texas
- Czechia (5):
  - Klecany
  - Litoměřice
  - Pilsen
  - Prague
  - Přerov
- Germany (12):
  - Berlin
  - Cham
  - Dresden
  - Gelsenkirchen
  - Halle
  - Leipzig
  - Mainz
  - Mannheim
  - Mittweida
  - Pfaffenhofen
  - Prien am Chiemsee
  - Tübingen
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Mysłowice
  - Pruszków
  - Torun
  - Tuszyn
  - Warsaw
- Spain (12):
  - Alcorcón
  - Barcelona
  - Córdoba
  - Málaga
  - Móstoles
  - Murcia
  - Palma
  - Pamplona
  - Sabadell
  - Salamanca
  - Santa Coloma de Gramanet
  - Vitoria-Gasteiz

REFERENCES:
- [Derived] Kaster TS, Dai Y, Vila-Rodriguez F, Downar J, Daskalakis ZJ, Blumberger DM, Rhee TG. Efficacy of intranasal esketamine versus rTMS for treatment-resistant depression: analysis of individual participant data from two clinical trials. EClinicalMedicine. 2025 Oct 30;90:103609. doi: 10.1016/j.eclinm.2025.103609. eCollection 2025 Dec. PMID 41245530
- [Derived] Kern Sliwa J, Naranjo RR Jr, Turkoz I, Petrillo MP, Cabrera P, Trivedi M. Effects of esketamine nasal spray on depressive symptom severity in adults with treatment-resistant depression and associations between the Montgomery-Asberg Depression Rating Scale and the 9-item Patient Health Questionnaire. CNS Spectr. 2024 Jun;29(3):176-186. doi: 10.1017/S1092852924000105. Epub 2024 Apr 1. PMID 38557430
- [Derived] Jamieson C, Popova V, Daly E, Cooper K, Drevets WC, Rozjabek HM, Singh J. Assessment of health-related quality of life and health status in patients with treatment-resistant depression treated with esketamine nasal spray plus an oral antidepressant. Health Qual Life Outcomes. 2023 May 8;21(1):40. doi: 10.1186/s12955-023-02113-1. PMID 37158911
- [Derived] Turkoz I, Nelson JC, Wilkinson ST, Borentain S, Macaluso M, Trivedi MH, Williamson D, Sheehan JJ, Salvadore G, Singh J, Daly E. Predictors of response and remission in patients with treatment-resistant depression: A post hoc pooled analysis of two acute trials of esketamine nasal spray. Psychiatry Res. 2023 May;323:115165. doi: 10.1016/j.psychres.2023.115165. Epub 2023 Mar 16. PMID 37019044
- [Derived] Jha MK, Williamson DJ, Magharehabed G, Turkoz I, Daly EJ, Trivedi MH. Intranasal esketamine effectively treats treatment-resistant depression in adults regardless of baseline irritability. J Affect Disord. 2023 Jan 15;321:153-160. doi: 10.1016/j.jad.2022.10.020. Epub 2022 Oct 20. PMID 36273682
- [Derived] Floden L, Hudgens S, Jamieson C, Popova V, Drevets WC, Cooper K, Singh J. Evaluation of Individual Items of the Patient Health Questionnaire (PHQ-9) and Montgomery-Asberg Depression Rating Scale (MADRS) in Adults with Treatment-Resistant Depression Treated with Esketamine Nasal Spray Combined with a New Oral Antidepressant. CNS Drugs. 2022 Jun;36(6):649-658. doi: 10.1007/s40263-022-00916-2. Epub 2022 Apr 20. PMID 35441931
- [Derived] Chen G, Chen L, Zhang Y, Li X, Lane R, Lim P, Daly EJ, Furey ML, Fedgchin M, Popova V, Singh JB, Drevets WC. Relationship Between Dissociation and Antidepressant Effects of Esketamine Nasal Spray in Patients With Treatment-Resistant Depression. Int J Neuropsychopharmacol. 2022 Apr 19;25(4):269-279. doi: 10.1093/ijnp/pyab084. PMID 35022754
- [Derived] Jones RR, Freeman MP, Kornstein SG, Cooper K, Daly EJ, Canuso CM, Nicholson S. Efficacy and safety of esketamine nasal spray by sex in patients with treatment-resistant depression: findings from short-term randomized, controlled trials. Arch Womens Ment Health. 2022 Apr;25(2):313-326. doi: 10.1007/s00737-021-01185-6. Epub 2022 Jan 1. PMID 34973081
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Daly EJ, Turkoz I, Salvadore G, Fedgchin M, Ionescu DF, Starr HL, Borentain S, Trivedi MH, Thase ME, Singh JB. The effect of esketamine in patients with treatment-resistant depression with and without comorbid anxiety symptoms or disorder. Depress Anxiety. 2021 Nov;38(11):1120-1130. doi: 10.1002/da.23193. Epub 2021 Jul 22. PMID 34293233
- [Derived] Turkoz I, Daly E, Singh J, Lin X, Tymofyeyev Y, Williamson D, Salvadore G, Nash AI, Macaluso M, Wilkinson ST, Nelson JC. Treatment Response With Esketamine Nasal Spray Plus an Oral Antidepressant in Patients With Treatment-Resistant Depression Without Evidence of Early Response: A Pooled Post Hoc Analysis of the TRANSFORM Studies. J Clin Psychiatry. 2021 Jul 20;82(4):20m13800. doi: 10.4088/JCP.20m13800. PMID 34288609
- [Derived] Doty RL, Popova V, Wylie C, Fedgchin M, Daly E, Janik A, Ochs-Ross R, Lane R, Lim P, Cooper K, Melkote R, Jamieson C, Singh J, Drevets WC. Effect of Esketamine Nasal Spray on Olfactory Function and Nasal Tolerability in Patients with Treatment-Resistant Depression: Results from Four Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase III Studies. CNS Drugs. 2021 Jul;35(7):781-794. doi: 10.1007/s40263-021-00826-9. Epub 2021 Jul 7. PMID 34235612
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208
- [Derived] Katz EG, Hough D, Doherty T, Lane R, Singh J, Levitan B. Benefit-Risk Assessment of Esketamine Nasal Spray vs. Placebo in Treatment-Resistant Depression. Clin Pharmacol Ther. 2021 Feb;109(2):536-546. doi: 10.1002/cpt.2024. Epub 2020 Oct 13. PMID 32860422
- [Derived] Saad Z, Hibar D, Fedgchin M, Popova V, Furey ML, Singh JB, Kolb H, Drevets WC, Chen G. Effects of Mu-Opiate Receptor Gene Polymorphism rs1799971 (A118G) on the Antidepressant and Dissociation Responses in Esketamine Nasal Spray Clinical Trials. Int J Neuropsychopharmacol. 2020 Dec 3;23(9):549-558. doi: 10.1093/ijnp/pyaa030. PMID 32367114
- [Derived] Popova V, Daly EJ, Trivedi M, Cooper K, Lane R, Lim P, Mazzucco C, Hough D, Thase ME, Shelton RC, Molero P, Vieta E, Bajbouj M, Manji H, Drevets WC, Singh JB. Efficacy and Safety of Flexibly Dosed Esketamine Nasal Spray Combined With a Newly Initiated Oral Antidepressant in Treatment-Resistant Depression: A Randomized Double-Blind Active-Controlled Study. Am J Psychiatry. 2019 Jun 1;176(6):428-438. doi: 10.1176/appi.ajp.2019.19020172. Epub 2019 May 21. PMID 31109201
- See also: A Randomized, Double-blind, Multicenter, Active-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Flexible Doses of Intranasal Esketamine Plus an Oral Antidepressant in Adult Subjects with Treatment-resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107147&attachmentIdentifier=512d9c31-6ce0-4e92-b568-a7ef54a494d2&fileName=ESKETINTRD3002_(CR107147)_Additional_results_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 236 participants were enrolled, out of which 227 were randomized and 9 participants were excluded due to Good Clinical Practice (GCP) violations.
Groups:
- Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD): Participants self-administered (under direct supervision by HCP) esketamine 56 milligram (mg) or 84 mg intranasally twice weekly for 4 weeks (on Day 1,4,8,11,15,18,22,25). Simultaneously, participants initiated per fixed titration scheme a new open-label oral AD with one of following: [Duloxetine (60 milligram (mg)/day- Weeks 1-4 with minimum dose for tolerability [MDT] of 60 mg/day); Escitalopram (10 mg/day-Week 1 and 20 mg/day- Weeks 2-4 with MDT of 10 mg/day); Sertraline (50 mg/day-Week 1, 100 mg/day-Week 2, 150 mg/day-Week 3 and 200 mg/day-Week 4 with MDT of 50 mg/day) or Venlafaxine XR (75 mg/day-Week 1, 150 mg/day-Week 2, and 225 mg/day-Weeks 3 and 4 with MDT of 150 mg/day) during DB Induction Phase. Participants who were not eligible or who chose to not participate in maintenance of effect study (ESKETINTRD3003[NCT02493868]) and had received at least 1 dose of intranasal Esketamine+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks.
- Intranasal Placebo Plus Oral AD: Participants self-administered (under direct supervision by HCP) esketamine matched placebo intranasally twice weekly for 4 weeks (on Day 1,4,8,11,15,18,22 and 25). Simultaneously, participants initiated per fixed titration scheme a new open-label oral AD with one of following: [Duloxetine (60 milligram (mg)/day- Weeks 1-4 with minimum dose for tolerability [MDT] of 60 mg/day); Escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2-4 with MDT of 10 mg/day); Sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MDT of 50 mg/day) or Venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, and 225 mg/day- Weeks 3 and 4 with MDT of 150 mg/day) during DB Induction Phase. Participants who were not eligible or who chose to not participate in maintenance of effect study (ESKETINTRD3003 [NCT02493868]) and had received at least 1 dose of intranasal Placebo+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks.
Period: Double Blind (DB) Phase (4 Weeks)
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Started | 116 | 111
Safety Analysis Set | 115 | 109
Full Analysis Set | 114 | 109
Completed | 98 | 99
Not Completed | 18 | 12
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Lack of Efficacy | 2 | 0
Not completed — Adverse Event | 9 | 1
Not completed — Other | 0 | 1
Period: Follow-up Phase (24 Weeks)
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Started | 34 | 52
Completed | 16 | 27
Not Completed | 18 | 25
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Investigator Decision | 6 | 17
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least 1 dose of intranasal study medication or
  1 dose of oral antidepressant medication during the double-blind induction phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD | Total
Number analyzed (Participants) | 115 | 109 | 224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 115 | 109 | 224
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12.56) | 46.4 (11.14) | 45.7 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 63 | 139
  Male | 39 | 46 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 109 | 99 | 208
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 107 | 102 | 209
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  CZECH REPUBLIC | 30 | 28 | 58
  GERMANY | 10 | 10 | 20
  POLAND | 20 | 18 | 38
  SPAIN | 9 | 9 | 18
  UNITED STATES | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score up to Day 28 in the Double-blind Induction Phase- Mixed-Effects Model Using Repeated Measures (MMRM) Analysis
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition.
Time Frame: Baseline up to Day 28 of Double-blind Induction Phase
Population: Full analysis set (FAS) defined as all randomized participants who received at least 1 dose of intranasal study medication, 1 dose of oral antidepressant (AD) medication during double-blind induction phase (D-BIP). Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 101 | 100
Units on a scale | -21.4 (12.32) | -17.0 (13.88)
Statistical Analysis 1: Comparison: Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) vs Intranasal Placebo Plus Oral AD; Test type: Superiority; p = 0.020, Mixed Model for Repeated Measures; Difference of Least Square (LS) Means = -4.0, 95% CI 2-sided [-7.31 to -0.64], Standard Error of Mean 1.69

2. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- Analysis of Covariance (ANCOVA) Analysis
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Endpoint (Double-blind Induction Phase [Day 28])
Population: FAS defined as all randomized participants who received at least 1 dose of intranasal study medication, 1 dose of AD medication during double-blind induction phase (D-BIP). Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 112 | 109
Units on a scale | -19.6 (13.58) | -16.3 (14.24)
Statistical Analysis 1: Comparison: Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) vs Intranasal Placebo Plus Oral AD; Test type: Superiority; p = 0.034, ANCOVA; Difference of Least Square (LS) Means = -3.5, 95% CI 2-sided [-6.67 to -0.26]

3. Secondary Outcome: Percentage of Participants With Onset of Clinical Response on Day 2 and Day 8
Description: A participant was defined as having a clinical response if there is at least 50 percent (%) improvement from baseline in the MADRS total score with onset by Day 2 and Day 8 that was maintained to Day 28. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. Participants who did not meet such criterion or discontinue during the study before Day 28 for any reason were considered as non-responders.
Time Frame: Day 2 up to Day 28 and Day 8 up to Day 28
Population: FAS is defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during the double-blind induction phase.
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 114 | 109
Percentage of participants
  Onset of Clinical response on Day 2 | 7.9 | 4.6
  Onset of Clinical response on Day 8 | 10.5 | 6.4

4. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score up to Day 28 of Double-blind Induction Phase- MMRM Analysis
Description: The SDS is a participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. First three items assess disruption of 1 work/school, 2 social life, 3 family life/home responsibilities using a 0(no impairment)-10 (most severe impairment). Score for first 3 items are summed to create total score of 0-30 where higher score indicates greater impairment and a negative change in score indicates improvement. It also has one item on days lost from school or work and one item on days when under productive.
Time Frame: Baseline up to Day 28 of Double-blind Induction phase
Population: FAS is defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during double-blind induction phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 86 | 85
Units on a scale | -13.6 (8.31) | -9.4 (8.43)

5. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis
Description: The SDS is a participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. First three items assess disruption of 1 work/school, 2 social life, 3 family life/home responsibilities using a 0(no impairment)-10 (most severe impairment). Score for first 3 items are summed to create total score of 0-30 where higher score indicates greater impairment and a negative change in score indicates improvement. It also has one item on days lost from school or work and one item on days when under productive. The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 95 | 89
Units on a scale | -12.5 (8.85) | -9.3 (8.39)

6. Secondary Outcome: Change From Baseline in Patient Health Questionnaire - 9-Item Depression Module (PHQ-9) Total Score up to Day 28 of Double-blind Induction Phase- MMRM Analysis
Description: PHQ-9 is 9-item, self-report scale assessing depressive symptoms. Each item is rated on 4-point scale (0=Not at all, 1=Several Days, 2=More than half days, 3=Nearly every day. Scale scores each of 9 symptom domains of Diagnostic and Statistical Manual of Mental Disorders, Major Depressive Disorder criteria and it has been used both as screening tool and measure of response to treatment for depression. The participant's item responses are summed to provide a total score (range of 0 to 27) with higher scores indicating greater severity of depressive symptoms. Severity of PHQ-9 categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19), Severe (20-27).
Time Frame: Baseline up to Day 28 of Double-blind Induction phase
Population: FAS is defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during double-blind induction phase. Here 'N' signifies overall number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 104 | 100
Units on a scale | -13.0 (6.42) | -10.2 (7.80)

7. Secondary Outcome: Change From Baseline in Patient Health Questionnaire - 9-Item Depression Module (PHQ-9) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])- ANCOVA Analysis
Description: PHQ-9 is 9-item, self-report scale assessing depressive symptoms. Each item is rated on 4-point scale (0=Not at all, 1=Several Days, 2=More than half days, 3=Nearly every day). Scale scores each of 9 symptom domains of Diagnostic and Statistical Manual of Mental Disorders, Major Depressive Disorder criteria and it has been used both as screening tool and measure of response to treatment for depression. The participant's item responses are summed to provide a total score (range of 0 to 27) with higher scores indicating greater severity of depressive symptoms. Severity of PHQ-9 categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19), Severe (20-27). The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 111 | 105
Units on a scale | -12.2 (6.87) | -10.1 (7.87)

8. Secondary Outcome: Percentage of Participants Who Achieved >=50% Reduction From Baseline in MADRS Total Score at the Endpoint (Double-blind Induction Phase [Day 28])
Description: MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. The percentage of participants with greater than or equal to (>=) 50 % reduction from baseline in MADRS total score was reported. The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: At Endpoint (Double-blind Induction Phase [Day 28])
Population: FAS is defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during the double-blind induction phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 112 | 109
Percentage of participants | 63.4 | 49.5

9. Secondary Outcome: Percentage of Participants in Remission (MADRS<=12) at the Endpoint (Double-blind Induction Phase [Day 28])
Description: Remission was defined as participants who had a MADRS total score of less than or equal to (=<) 12. MADRS is clinician-rated scale designed to measure depression severity, and to detect changes due to antidepressant treatment. Scale consists of 10 items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts), each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of symptoms), summed for a total possible score of 0 to 60. Higher scores represent more severe condition. The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: At Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 112 | 109
Percentage of participants | 48.2 | 30.3

10. Secondary Outcome: Percentage of Participants in Response (SDS Total Score <=12 and Individual Item Scores Each <=4) at the End of 4-Week Double-blind Induction Phase (Day 28)
Description: Response defined as SDS total score <= 12 and individual item scores each <= 4. SDS is a participant-reported outcome measure and 5 item questionnaire used for assessment of functional impairment and associated disability. First three items assess disruption of 1 work/school, 2 social life, 3 family life/home responsibilities using a 0(no impairment)-10 (most severe impairment). Score for first 3 items are summed to create total score of 0-30 where higher score indicates greater impairment and a negative change in score indicates improvement. It also has one item on days lost from school or work and one item on days when under productive.
Time Frame: At Day 28 [end of Double-blind Induction Phase]
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 86 | 86
Percentage of participants | 57.0 | 39.5

11. Secondary Outcome: Percentage of Participants in Remission (SDS Total Score <=6 and Individual Item Scores Each <=2) at the End of 4-Week Double-blind Induction Phase (Day 28)
Description: Remission defined as SDS total score <= 6 and individual item scores each <= 2. SDS is a participant reported outcome measure and is a 5-item questionnaire which has been widely used and accepted for assessment of functional impairment and associated disability. The first three items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a 0-10 rating scale. The score for the first three items were summed to create a total score of 0-30 where a higher score indicates greater impairment. It also has one item on days lost from school or work and one item on days when under productive.
Time Frame: At Day 28 (End of Double-blind Induction Phase)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 86 | 86
Percentage of participants | 39.5 | 20.9

12. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])
Description: CGI-S provides measure of severity of participant's illness including participant's history, psychosocial circumstances, symptoms, behavior and impact of symptoms on ability to function. CGI-S evaluates severity of psychopathology on scale of 0 to 7. Considering total clinical experience, participant is assessed on severity of mental illness according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among most extremely ill patients. CGI-S permits global evaluation of participant's condition at given time. The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Endpoint (Double-blind Induction Phase [Day 28])
Population: FAS defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during the double-blind induction phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 111 | 109
Units on a scale | -2.0 [-5 to 1] | -2.0 [-5 to 1]

13. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder (GAD-7) Total Score up to Endpoint (Double-blind Induction Phase [Day 28])
Description: GAD-7 is a brief and validated 7-item self-report assessment of overall anxiety. Participants respond to each item using a 4-point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score with a range of 0 to 21, where higher scores indicate more anxiety. The recall period is 2 weeks. The severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14) and Severe (15 -21). The last post baseline observation during the phase was carried forward as "End Point" for that phase.
Time Frame: Baseline up to Endpoint (Double-blind Induction Phase [Day 28])
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 110 | 102
Units on a scale | -7.9 (6.12) | -6.8 (5.75)

14. Secondary Outcome: Change From Baseline in EQ 5D-5L-Health Status Index to End of Double-blind Induction Phase (Day 28)
Description: European Quality of Life Group-5 Dimension-5-Level (EQ-5D-5L) is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). Health Status Index range is -0.148 - 0.949, is anchored at 0 (dead) and 1 (full health).
Time Frame: Baseline up to End of Double-blind Induction Phase (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 111 | 105
Units on a Scale | 0.288 (0.2317) | 0.231 (0.2506)

15. Secondary Outcome: Change From Baseline in EQ 5D-5L- European Quality of Life - Visual Analogue Scale (EQ-VAS) to End of Double-blind Induction Phase (Day 28)
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Time Frame: Baseline up to End of Double-blind Induction Phase (Day 28)
Population: FAS is defined as all randomized participants who received at least 1 dose of intranasal study medication and 1 dose of oral AD medication during the double blind induction phase. Here 'N' (overall number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 111 | 105
Units on a scale | 29.1 (26.32) | 20.9 (26.60)

16. Secondary Outcome: Change From Baseline in EQ 5D-5L- Sum Score to End of Double-blind Induction Phase (Day 28)
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ VAS). EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). Health Status Index range is -0.148 - 0.949, is anchored at 0 (dead) and 1 (full health). EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline up to End of Double-blind Induction Phase (Day 28)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intranasal Esketamine (Esk) Plus Oral Antidepressant (AD) | Intranasal Placebo Plus Oral AD
Number analyzed (Participants) | 111 | 105
Units on a scale | -23.2 (16.64) | -17.1 (19.66)

ADVERSE EVENTS:
Time Frame: Approximately up to 2.2 Years
Description: The safety analysis set included all randomized participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant medication during the double-blind induction phase. The follow-up analysis set included all participants who entered the follow-up phase.
Groups:
- DB Phase: Intranasal Esk + Oral AD: Participants self-administered (under direct supervision by health care professional [HCP]) esketamine either 56 milligram (mg) or 84 mg intranasally twice weekly for 4 weeks (on Day 1, 4, 8, 11, 15, 18, 22 and 25). Simultaneously, participants initiated per fixed titration scheme a new open-label oral antidepressant (AD) with one of following: [Duloxetine (60 milligram (mg)/day- Weeks 1-4 with minimum dose for tolerability [MDT] of 60 mg/day); Escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2-4 with MDT of 10 mg/day); Sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MDT of 50 mg/day) or Venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, and 225 mg/day- Weeks 3 and 4 with MDT of 150 mg/day) during DB Induction Phase.
- DB Phase: Oral AD + Intranasal Placebo: Participants self-administered (under direct supervision by HCP) esketamine matched placebo intranasally twice weekly for 4 weeks (on Day 1, 4, 8, 11, 15, 18, 22 and 25). Simultaneously, participants initiated per fixed titration scheme a new open-label oral AD with one of following: [Duloxetine (60 milligram (mg)/day- Weeks 1-4 with minimum dose for tolerability [MDT] of 60 mg/day); Escitalopram (10 mg/day- Week 1 and 20 mg/day- Weeks 2-4 with MDT of 10 mg/day); Sertraline (50 mg/day- Week 1, 100 mg/day- Week 2, 150 mg/day- Week 3 and 200 mg/day- Week 4 with MDT of 50 mg/day) or Venlafaxine XR (75 mg/day- Week 1, 150 mg/day- Week 2, and 225 mg/day- Weeks 3 and 4 with MDT of 150 mg/day) during DB Induction Phase.
- FU Phase: Intranasal Esk + Oral AD: Participants who were not eligible or who chose to not participate in maintenance of effect study (ESKETINTRD3003 [NCT02493868]) and had received at least 1 dose of intranasal Esk+ Oral AD in DB induction phase were followed in posttreatment follow-up (FU) phase for up to 24 weeks.
- FU Phase: Oral AD + Intranasal Placebo: Participants who were not eligible or who chose to not participate in maintenance of effect study (ESKETINTRD3003 [NCT02493868]) and had received at least 1 dose of intranasal Placebo+ Oral AD in DB induction phase were followed in posttreatment follow-up phase for up to 24 weeks.
Arm/Group | DB Phase: Intranasal Esk + Oral AD | DB Phase: Oral AD + Intranasal Placebo | FU Phase: Intranasal Esk + Oral AD | FU Phase: Oral AD + Intranasal Placebo
All-Cause Mortality (participants affected / at risk) | 1/115 | 0/109 | 0/34 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/115 | 1/109 | 1/34 | 0/52
Other Adverse Events (participants affected / at risk) | 90/115 | 53/109 | 7/34 | 6/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Intranasal Esk + Oral AD (N=115) | DB Phase: Oral AD + Intranasal Placebo (N=109) | FU Phase: Intranasal Esk + Oral AD (N=34) | FU Phase: Oral AD + Intranasal Placebo (N=52)
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Phase: Intranasal Esk + Oral AD (N=115) | DB Phase: Oral AD + Intranasal Placebo (N=109) | FU Phase: Intranasal Esk + Oral AD (N=34) | FU Phase: Oral AD + Intranasal Placebo (N=52)
Vertigo (Ear and labyrinth disorders) | 30 | 3 | 0 | 0
Vision Blurred (Eye disorders) | 14 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 10 | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 9 | 3 | 1 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 9 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 30 | 7 | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 9 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 2 | 0 | 0
Fatigue (General disorders) | 5 | 6 | 0 | 0
Feeling Drunk (General disorders) | 9 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 3 | 0
Blood Pressure Increased (Investigations) | 11 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0
Dizziness (Nervous system disorders) | 24 | 5 | 1 | 2
Dizziness Postural (Nervous system disorders) | 8 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 28 | 13 | 0 | 0
Headache (Nervous system disorders) | 23 | 19 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 8 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 13 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 15 | 7 | 0 | 0
Anxiety (Psychiatric disorders) | 12 | 5 | 1 | 1
Dissociation (Psychiatric disorders) | 30 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 5 | 0 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 0 | 0

LIMITATIONS AND CAVEATS:
As this was a flexible-dose study, dose-response relationships could not be evaluated because direct comparisons between dose groups could not be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02418585/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02418585/SAP_001.pdf